CLINICAL TRIAL: NCT03349970
Title: Intraoperative Measurement of Cardiac Output During Cardiac Surgery: Which TEE Method is Best?
Brief Title: Cardiac Output Measurement by TEE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jo Carroll, Research Manager, University Health Network, Toronto
Other Study IDs: 16-6341
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TEE vs PAC: we will compare the SV measurements obtained by PAC thermodilution technique to those obtained by different TEE methods in 60 patients undergoing coronary artery bypass grafting (CABG) and/or aortic valve (AV) or aortic surgery with cardiopulmonary bypass (CPB) in 2 different cardiac centres. The LV cardiac deformation, expressed as global longitudinal strain (GLS) will be calculated off-line from the acquired images. We will also determine the intra and inter-observer reproducibility of each TEE method.

SUMMARY:
Transesophageal echocardiography (TEE) has become a standard monitoring tool during cardiac surgery. It allows continuous accurate assessment of heart structures and function without interfering with the surgery and the anesthetics. The imaging of cardiac structures is used to direct optimal surgical intervention and assess surgical results. Cardiac output (CO) is the result of stroke volume (SV) multiplied by the heart rate.

Measurement of cardiac output (CO) is used to quantify the performance of the left ventricle. It is commonly achieved using a pulmonary artery catheter (PAC) (also known ad Swann-Ganz catheter). A known amount of saline solution is injected in the proximal part of the catheter and the variation of blood temperature detected at the tip. Cardiac output is measured based on the duration and degree of temperature change. This method remains an accepted gold standard. TEE allows measurement of cardiac output using a number of different 2D and 3D imaging modalities. Although current guidelines identify the Method of the Disks(MOD) as the gold standard other technique could potentially be more precise. In this study, the investigators want to assess the accuracy of four different TEE methods to measure cardiac output compared with Thermodilution as a standard of care.

DETAILED DESCRIPTION:
The measurement of the LV performance, as reflected by measuring cardiac output (CO), is an important component of hemodynamic assessment during cardiac (and non-cardiac) surgery. It has become standard of care in guiding fluid management and inotropic therapy in both the operating room (OR) and the intensive care unit (ICU) in most centres, and is considered by far the most understood and commonly communicated parameter of cardiac performance, in addition to being consistently shown as a predictor of patients' outcome.

Several methods have been used to measure CO. The most commonly used is via thermodilution (PAC), but its invasive nature and potential for serious complications led to the utilization of the non-invasive methods, such as those based on TEE.

Since the establishment of the role of TEE in the setting of hemodynamic monitoring during cardiac surgery, various ways of quantifying LV function have been utilized. The method recommended by current guidelines is a volumetric calculation via the method of disks (modified Simpson's method, MOD). Recent advances in ultrasound technology and software development allow the utilization three-dimensional (3D) volumetric assessment and speckle tracking for cardiac deformation.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* undergoing elective CABG, AV or aortic surgery (aortic root and ascending aortic arch surgery), with CPB.

Exclusion Criteria:

* Emergency surgery
* Moderate or severe valve pathology
* Atrial fibrillation
* Patients with known contraindications to either the insertion of a PAC or the use of TEE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac patients undergoing elective CABG, AV or aortic surgery (aortic root and ascending aortic arch surgery), with CPB
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
The primary Objective is to compare five different intraoperative echocardiographic measurements of cardiac output with the gold standard thermodilution in patients undergoing elective cardiac surgery. | Intraoperatively

SECONDARY OUTCOMES:
The secondary objective is to test each TEE method against the standard of care method of the disks | Intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Meineri, MD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Weill Cornell Medicine, New York, New York, United States
- Toronto General Hopsital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No